CLINICAL TRIAL: NCT03028428
Title: Clinical Research on Intra-articular Injection of Human Autologous MSCs in Treatment of Knee OA
Brief Title: Intra-articular Injection of MSCs in Treatment of Knee OA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Affiliated Hospital of Jiangsu University (Other)
Responsible Party: Principal Investigator, YU TANG, Dr., Affiliated Hospital of Jiangsu University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHJiangsuU-FSK-MSC-OA
Record Dates: First submitted 2017-01-20; First posted 2017-01-23 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis; Stem Cells; MSC
Keywords: Osteoarthritis; Stem Cell; Knee; Mesenchymal Stem Cell
MeSH Terms: conditions — Osteoarthritis | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: A Randomized, Double Blind, Phase-II Study Assessing the Safety and Efficacy of Intraarticular Ex-vivo Cultured Adult Allogeneic Mesenchymal Stem Cells in Patients with Osteoarthritis of Knee
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind

ARMS (2):
- Placenta Derived Mesenchymal Stem Cell (Experimental): Placenta Derived Mesenchymal Stem Cell administered into the knee joint once
  Interventions: Biological: Placenta Derived Mesenchymal Stem Cell
- sodium hyaluronate (Active Comparator): Sodium hyaluronate administered into the knee joint once
  Interventions: Drug: Sodium Hyaluronate

INTERVENTIONS:
Biological: Placenta Derived Mesenchymal Stem Cell — 1ml 1*10^7 Placenta Derived Mesenchymal Stem Cell administered into the knee joint once
  Other Names: Mesenchymal Stromal Cells (MSCs)
  Arms: Placenta Derived Mesenchymal Stem Cell
Drug: Sodium Hyaluronate — Sodium hyaluronate administered into the knee joint once
  Other Names: hyaluronate
  Arms: sodium hyaluronate

SUMMARY:
In this study, researchers want to determine the safety of MSCs that a patient can tolerate without causing side effects. Moreover researchers will also be looking at the function of the knee over time, which may give them some insight on the usefulness of MSCs as a treatment option.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most common forms of arthritis. It is a lasting condition in which the material that cushions the joints, called cartilage, breaks down. This causes the bones to rub against each other, causing inflammation, stiffness, pain and loss of joint movement. Currently, there are few effective treatments available for patients suffering from OA.

Mesenchymal stem cells (MSCs) are cells that have the ability to self-regenerate, which means they have the ability to make copies of themselves and to turn into other kinds of cells (e.g. cartilage cells). Stem cell science shows much promise for the future treatment of osteoarthritis, but much of the research is still in the early stages. In this study, researchers want to determine the safety of MSCs that a patient can tolerate without causing side effects. Moreover researchers will also be looking at the function of the knee over time, which may give them some insight on the usefulness of MSCs as a treatment option.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 40-75 years of age with symptomatic moderate to severe (Kellgren-Lawrence III or IV) primary osteoarthritis of the knee
2. Idiopathic or secondary osteoarthritis of the knee with grade 2,3, or 4 radiographic severity, as defined by the modified Kellgren-Lawrence classification
3. No history of prior intra-articular cortisone, hyaluronic acid, or platelet-rich plasma injection within the previous six months
4. No history of prior arthroscopic knee surgery or open knee surgery on the ipsilateral side within the past year
5. Adequate bone marrow, liver, and renal functions
6. Body weight >40 kg
7. Body Mass Index <40
8. Negative for (HIV, HTLV1&2, Hep A, B, C, syphilis) infection as determined by approved serological testing
9. Negative for pregnancy as determined by a serum pregnancy test. Females of childbearing potential will be required to practice abstinence or use an effective form of contraception for 12 months following their MSC injection.
10. Ability to provide written informed consent.

Exclusion Criteria:

1. Patients with clinically unstable knee due to the presence of a complete anterior cruciate ligament, posterior cruciate ligament, medial collateral ligament and/or posterolateral corner tear
2. Patients with varus or valgus malalignment >5 degrees as measured by 4 foot standing antero-posterior radiographs
3. Patients with a history of a previous subtotal medial or lateral meniscectomy
4. Patients with a history of septic arthritis in the affected joint
5. Patients with a history of a prior intra-articular knee fracture
6. Severe bleeding diathesis
7. Contraindication to bone marrow aspiration and/or biopsy
8. Active infection
9. Bone marrow failure
10. Cytopenia
11. Patients who have previously received radiotherapy to the pelvis
12. Patients who have been on chemotherapy from within a year of the date of informed
13. Patients with positive serological test for (HIV, HTLV1&2, Hep A, B, C, syphilis)
14. Pregnancy or risk of pregnancy (this includes participants that are not willing to practice active contraception for the duration of the study)
15. Patients with unforeseen conditions that are deemed unsafe or inappropriate for the study (e.g. patients who are claustrophobic and cannot undergo an MRI) as per the discretion of the principal investigator

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
adverse events | 1 Year
  Number of participants with adverse events as measure of safety and tolerability

SECONDARY OUTCOMES:
radiographic evidence | 1 Year
  Number of participants with a change in cartilage thickness of knee OA using MRI
WOMAC assessment | 1 Year
  Number of participants with a change in joint function from baseline WOMAC assessment
VAS | 1 Year
  Number of participants with a change in arthritis pain scores on the visual analogue scale
SF-36 | 1 Year
  Number of participants with a change in SF-36

CONTACTS AND LOCATIONS:
Overall Officials: YU TANG, Dr., Principal Investigator — Affiliated Hospital of Jiangsu University